CLINICAL TRIAL: NCT01009190
Title: A Parallel Arms Phase 1 Safety, Pharmacokinetic And Pharmacodynamic Study Of The Intravenous Poly (ADP-Ribose) Polymerase (PARP) Inhibitor PF-01367338 (AG-014699) In Combination With Several Chemotherapeutic Regimens In Adult Patients With Advanced Solid Tumor
Brief Title: A Study Of Poly (ADP-Ribose) Polymerase Inhibitor PF-01367338 In Combination With Several Chemotherapeutic Regimens
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-1014
Record Dates: First submitted 2009-11-04; First posted 2009-11-06 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumors
Keywords: Dose finding PARPi Chemotherapy
MeSH Terms: interventions — rucaparib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Experimental): Carboplatin plus PF-01367338
  Interventions: Drug: PF-01367338; Drug: Carboplatin
- ARM A EXPANSION (Experimental): Carboplatin plus PF-01367338
  Interventions: Drug: PF-01367338; Drug: Carboplatin

INTERVENTIONS:
Drug: PF-01367338 — Increasing doses of single lead-in (Day -10) intravenous and daily oral PF-01367338 administered from Day 1 to Day 14 every 3-week cycle
  Arms: ARM A
Drug: Carboplatin — Standard doses of intravenous Carboplatin administered every 3 weeks
  Arms: ARM A
Drug: PF-01367338 — RP2 doses of oral PF-01367338 administered daily from Day 1 to Day 14 every 3-week cycle
  Arms: ARM A EXPANSION
Drug: Carboplatin — Standard doses of intravenous Carboplatin administered every 3 weeks
  Arms: ARM A EXPANSION

SUMMARY:
Dose escalation phase 1 study of PARP inhibitor PF-01367338 in combination with chemotherapy in adult patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed solid tumors, Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Patients with acceptable renal, hepatic, and bone marrow function

Exclusion Criteria:

* Symptomatic and/or unstable brain metastases,
* Any cancer treatment within 4 weeks from study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of escalating doses of PF-01367338 in combination with chemotherapy (as defined by first-cycle DLTs) | 18 months
  Dose-limiting toxicities and adverse events

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics of escalating doses of PF-01367338 in combination with several chemotherapeutic regimens | 18 months
  Time to attain maximum plasma concentration [Tmax]
Pharmacokinetics and pharmacodynamics of escalating doses of PF-01367338 in combination with several chemotherapeutic regimens | 18 months
  maximum plasma concentration (CMax)
Pharmacokinetics and pharmacodynamics of escalating doses of PF-01367338 in combination with several chemotherapeutic regimens | 18 months
  area under plasma concentration curve (AUC)
Pharmacokinetics and pharmacodynamics of escalating doses of PF-01367338 in combination with several chemotherapeutic regimens | 18 months
  apparent terminal half-life (t1/2)
Pharmacokinetics and pharmacodynamics of escalating doses of PF-01367338 in combination with several chemotherapeutic regimens | 18 months
  rucaparib oral bioavailability
PARP activity and expression in peripheral blood lymphocytes (PBL) | 18 months
  % PARP activity
Determination of food effect on oral PF-01367338 pharmacokinetics | 18 month
  fasted and fed parameters area under the plasma concentration-time curve from time 0 to the last recorded observation [AUClast]
Determination of food effect on oral PF-01367338 pharmacokinetics | 18 month
  fasted and fed maximum plasma concentration (Cmax)
Determination of effect of PF-013567338 administration on QTc prolongation test | 18 months
  electrocardiogram[ecg], QTcF, QTcB

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Churchill Hospital, Oxford, Oxfordshire
  - Royal Marsden Hospital, Sutton, Surrey
  - Belfast City Hospital, Belfast
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Kings College London, London
  - Sir Bobby Robson Cancer Trials Research Centre, Newcastle upon Tyne

REFERENCES:
- [Derived] Green ML, Ma SC, Goble S, Giordano H, Maloney L, Simmons AD, Beltman J, Harding TC, Xiao JJ. Population pharmacokinetics of rucaparib in patients with advanced ovarian cancer or other solid tumors. Cancer Chemother Pharmacol. 2022 May;89(5):671-682. doi: 10.1007/s00280-022-04413-7. Epub 2022 Apr 10. PMID 35397664
- [Derived] Wilson RH, Evans TJ, Middleton MR, Molife LR, Spicer J, Dieras V, Roxburgh P, Giordano H, Jaw-Tsai S, Goble S, Plummer R. A phase I study of intravenous and oral rucaparib in combination with chemotherapy in patients with advanced solid tumours. Br J Cancer. 2017 Mar 28;116(7):884-892. doi: 10.1038/bjc.2017.36. Epub 2017 Feb 21. PMID 28222073